CLINICAL TRIAL: NCT06230861
Title: Effects of Quercetin Supplementation on Cardiometabolic Parameters
Brief Title: Effects of Quercetin on Cardiometabolic Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Quercetin cardiometabolic
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-07

CONDITIONS: Cardiometabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quercetin tablets 400mg 1 x p/d (Experimental): Quercetin tablets 400mg 1 x p/d
  Interventions: Dietary Supplement: Quercetin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin — Quercetin tablets 500mg 1 x per day
  Arms: Quercetin tablets 400mg 1 x p/d
Other: Placebo — Placebo control 1 x blinded placebo tablet per day
  Arms: Placebo

SUMMARY:
Cardiovascular disease, type 2 diabetes mellitus and associated diseases combined are the leading health burden and cause of mortality worldwide; therefore, the necessity for an intervention is paramount. Dietary interventions to improve cardiometabolic health are highly sought after as they possess less risk than pharmacological drugs. It has been postulated that Quercetin may be beneficial in improving cardiometabolic outcomes. However, to date, no research has explored this using a placebo randomized intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Between 18 & 65 years
* Non-smoker
* BMI < 30
* Able to give informed consent

Exclusion Criteria:

* Pregnancy
* Diabetes or any other metabolic/ uncontrolled hypertensive conditions
* Food allergies to quercetin
* Habitual consumption of quercetin
* Not regularly taking medication or antioxidant supplements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline
  Systolic blood pressure - measured using a digital blood pressure monitor
Systolic blood pressure | 20 days
  Systolic blood pressure - measured using a digital blood pressure monitor

SECONDARY OUTCOMES:
Diastolic blood pressure | Baseline
  Diastolic blood pressure - measured using a digital blood pressure monitor
Diastolic blood pressure | 20 days
  Diastolic blood pressure - measured using a digital blood pressure monitor
Percent bodyfat | Baseline
  Participants percentage composition of fat - measured using bio-electrical impedance
Percent bodyfat | 20 days
  Participants percentage composition of fat - measured using bio-electrical impedance
Waist to hip ratio | Baseline
  Ratio of waist to hip circumference - measured using anthropocentric tape
Waist to hip ratio | 20 days
  Ratio of waist to hip circumference - measured using anthropocentric tape
Blood glucose | Baseline
  Capillary blood glucose - mmol/L
Blood glucose | 20 days
  Capillary blood glucose - mmol/L
Blood triglycerides | Baseline
  Capillary blood triglycerides - mmol/L
Blood triglycerides | 20 days
  Capillary blood triglycerides - mmol/L
Triglyceride glucose index | Baseline
  Calculated as the natural logarithm of (blood triglycerides x blood glucose) /2)
Triglyceride glucose index | 20 days
  Calculated as the natural logarithm of (blood triglycerides x blood glucose) /2)
Blood cholesterol (Total, HDL & LDL) | Baseline
  Capillary blood cholesterol - mmol/L
Blood cholesterol (Total, HDL & LDL) | 20 days
  Capillary blood cholesterol - mmol/L
Coop-Wonka chart | Baseline
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring
Coop-Wonka chart | 20 days
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring
Beck Depression Inventory | Baseline
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Beck Depression Inventory | 20 days
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
State Trait Anxiety Inventory | Baseline
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
State Trait Anxiety Inventory | 20 days
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
Insomnia Severity Index | Baseline
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Insomnia Severity Index | 20 days
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Pittsburgh Sleep Quality Index | Baseline
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Pittsburgh Sleep Quality Index | 20 days
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Epworth Sleepiness Scale | Baseline
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Epworth Sleepiness Scale | 20 days
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No